CLINICAL TRIAL: NCT05462912
Title: Evaluation of Software Generated Customized Foot Orthoses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Per sponsor, trial criteria were not followed and the data collected is not available
Sponsor: University of California, Davis (Other)
Collaborators: Soleit (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1771535
Record Dates: First submitted 2022-04-27; First posted 2022-07-18 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Arthropathy of Ankle or Foot

STUDY DESIGN:
Intervention Model Description: Each participant will be evaluated at baseline, when the customized foot orthoses will be made, and the corresponding tests will be conducted
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Open (Other): Each participant will be evaluated at baseline, when the customized foot orthoses will be made, and the corresponding tests will be conducted.
  Interventions: Device: custom foot orthotic

INTERVENTIONS:
Device: custom foot orthotic — The goal of this study is to find out whether the use of software generated custom-made orthopedic foot orthoses improves pain in the long term.

SUMMARY:
The purpose of this study is to determine whether custom-made foot orthoses generate a significant decrease in the perception of pain among individuals with foot pain and/or ankle pain.

DETAILED DESCRIPTION:
The investigators aim to enroll up to 60 participants over the course of 1-3 months. Each participant will be evaluated at baseline, when the customized foot orthoses will be made, and the corresponding tests will be conducted. Subsequently, consecutive surveys will be carried out at 0, 7, 30, 120, and 360 days from the first day of foot orthoses use to measure the change in pain and comfort with use of the foot orthoses. An interim analysis will be conducted after all subjects have completed the 30-day time point. This interim analysis will allow the sponsor to determine whether subjects are using the foot orthoses that the subjects have been provided. Complete primary analysis is estimated to be completed within 3 months after the termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Foot/ankle pain or pathology OR diagnosed pes planus, pes cavus, pronator foot, supinator foot, metatarsalgia, Morton's neuroma, sesamoiditis, hallux valgus, intermetatarsal bursitis
2. Between 18 and 65 years of age
3. BMI is greater than 18.5 or less than 30

Exclusion Criteria:

1. Individuals who have had surgery in the lower limbs during this past year.
2. Individuals who already have custom-made orthopedic orthoses.
3. Patients with active diabetic ulcers or chronic foot pressure ulcers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Giza, MD, Principal Investigator — UC Davis Orthopaedic Surgery
Locations (1):
- UC Davis Health, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Open
Started | 60
Completed (Trial terminated due to sponsor decision.) | 0
Not Completed | 60

BASELINE CHARACTERISTICS:
Population: Subjects complaining of foot pain.
Arm/Group | Open
Number analyzed (Participants) | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 45 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 60
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Successful Patient Use of a 3D Printed Custom Foot Orthotic
Description: The purpose of this study is to determine whether custom-made foot orthoses generate a significant decrease in the perception of pain among individuals with foot pain and/or pathology.
  Secondary:
  1. To determine whether custom-made foot orthoses generate a significant increase in comfort among individuals with foot pain and/or pathology.
  2. To determine whether custom-made foot orthoses improve quality of life among individuals with foot pain and/or pathology
Time Frame: 11 months
Population: A random sampling of subjects presenting with the condition being studied
Measure: Number; unit: participants
Groups:
- Open: Each participant will be evaluated at baseline, when the customized foot orthoses will be made, and the corresponding tests will be conducted.
  custom foot orthotic: The goal of this study is to find out whether the use of software generated custom-made orthopedic foot orthoses improves pain in the long term.
  The purpose of this study is to determine whether custom-made foot orthoses generate a significant decrease in the perception of pain among individuals with foot pain and/or pathology.
  Secondary:
  1. To determine whether custom-made foot orthoses generate a significant increase in comfort among individuals with foot pain and/or pathology.
  2. To determine whether custom-made foot orthoses improve quality of life among individuals with foot pain and/or pathology.
Arm/Group | Open
Number analyzed (Participants) | 60
participants | 60

ADVERSE EVENTS:
Time Frame: 11 months after completion of screening visit.
Description: Because this study is subjective in nature, only adverse events that are serious, unexpected, and device-related will be recorded. Collection of adverse events will begin once subject begins using the foot orthoses. All adverse events will be monitored and reported in accordance with the UC Davis Institutional Review Board (IRB) policies
Groups:
- Open: Each participant will be evaluated at baseline, when the customized foot orthoses will be made, and the corresponding tests will be conducted.
  custom foot orthotic: The goal of this study is to find out whether the use of software generated custom-made orthopedic foot orthoses improves pain in the long term.
  Primary endpoint: Successful patient use of a 3D printed custom orthotic for at least 6 months and up to 1 year
Arm/Group | Open
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Due to significant issues identified in the data collection process the study was terminated prematurely The study required participants to complete a survey at three specific time points: This was not done.

The data was not stored and will not be used for any future analysis. No data was evaluated or stored that was collected for this trial. The website where data was originally collected was deleted and not accessible. No data analysis was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT05462912/Prot_000.pdf
  • Informed Consent Form (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/12/NCT05462912/ICF_001.pdf